CLINICAL TRIAL: NCT06932848
Title: The Therapeutic Effect of Curcumin in Nanogels Compared to 0.1% Fluocinolone Acetonide Oral Paste in the Management of Atrophic-Erosive Oral Lichen Planus
Brief Title: The Therapeutic Effect of Curcumin in Nanogels Compared to 0.1% FAO in the Management of Oral Lichen Planus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HREC-DCU 2025-007
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Oral Lichen Planus
Keywords: Atrophic-Erosive Oral Lichen Planus; Curcumin; Nanogels; Fluocinolone Acetonide; Mucosal Disease; Autoimmune Disease
MeSH Terms: conditions — Lichen Planus, Oral; Autoimmune Diseases | interventions — Curcumin; Nanogels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin Group (Experimental): Curcumin nanogels applied 3 times daily for 4 weeks
  Interventions: Drug: Curcumin in Nanogels
- Fluocinolone Paste Group (Active Comparator): 0.1% Fluocinolone acetonide oral paste applied 3 times daily for 4 weeks
  Interventions: Drug: 0.1% Fluocinolone Acetonide Oral Paste

INTERVENTIONS:
Drug: Curcumin in Nanogels — Participants will apply curcumin nanogels to affected oral areas three times daily for 4 weeks.
  Arms: Curcumin Group
Drug: 0.1% Fluocinolone Acetonide Oral Paste — Participants will apply 0.1% fluocinolone acetonide oral paste to the affected oral mucosa three times daily for 4 weeks. This corticosteroid paste is the standard treatment for oral lichen planus.
  Arms: Fluocinolone Paste Group

SUMMARY:
This randomized, double-blind clinical trial evaluates the therapeutic effects of curcumin in nanogels compared to 0.1% fluocinolone acetonide oral paste in the management of atrophic-erosive oral lichen planus (OLP). The study aims to determine whether curcumin nanogels, a natural treatment with enhanced bioavailability, are as effective and better tolerated than standard corticosteroid therapy.

DETAILED DESCRIPTION:
Oral lichen planus (OLP) is a chronic, immune-mediated inflammatory condition that causes painful mucosal lesions and significantly impairs patients' quality of life. Although topical corticosteroids are the standard treatment, their long-term use is associated with adverse effects. Curcumin, a natural compound with anti-inflammatory and antioxidant properties, has shown promise as an alternative treatment. However, its clinical application is limited by poor bioavailability.

This randomized, double-blind, controlled clinical trial aims to compare the therapeutic effects of curcumin in nanogels and 0.1% fluocinolone acetonide oral paste in patients with atrophic-erosive OLP. Thirty eligible participants will be randomly assigned to either the curcumin nanogel or fluocinolone group, and treatment outcomes will be evaluated using the Oral Lichen Planus Disease Activity Scale (OLP-DAS) and a patient satisfaction questionnaire over a 4-week period.

The study is conducted at the Faculty of Dentistry, Chulalongkorn University, and seeks to evaluate whether curcumin nanogels offer comparable therapeutic efficacy to corticosteroids, with potentially fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Ability to provide written informed consent
* Clinically and histopathologically confirmed diagnosis of erosive or atrophic oral lichen planus (OLP)
* Presence of symptoms (NRS pain score > 0 at baseline)
* Ability to communicate and follow instructions
* Willingness to apply oral paste treatment and comply with study protocol

Exclusion Criteria:

* Pregnancy or lactation
* Current orthodontic treatment
* Uncontrolled diabetes mellitus (HbA1c > 7% or FPG > 130 mg/dL)
* Use of anticoagulants or antiplatelet agents
* Severe dry mouth (Challacombe score > 7)
* History of gastric ulcers, duodenal ulcers, or gallstones
* Presence of any active malignancy or infection
* Use of topical/systemic treatment for OLP in the past 2 weeks
* Current use of immunosuppressants
* Known allergy to corticosteroids or herbal agents such as turmeric
* Diagnosis of oral lichenoid contact lesion or graft-versus-host disease (GVHD)
* History of allogeneic bone marrow transplantation
* Current smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in OLP-DAS Score | Baseline, 2 weeks, and 4 weeks
  Evaluation of change in Oral Lichen Planus-Disease Activity Scale (OLP-DAS) score, which includes lesion severity, lesion extent, and pain score, from baseline to follow-up
  The Oral Lichen Planus-Disease Activity Scale (OLP-DAS) includes 3 components:
  * OLP Sign Score (0-65)
  * OLP Severity Index (0-20)
  * Numerical Rating Scale for pain (0-10)
  The total OLP-DAS score ranges from 0 to 95. Higher scores indicate worse disease activity.

SECONDARY OUTCOMES:
Product Satisfaction Questionnaire | At 4 weeks after treatment start
  Product satisfaction will be evaluated using a modified 6-item Product Satisfaction Questionnaire. Items include:
  * Taste of the oral paste
  * Oral sensation
  * Irritation
  * Convenience of use
  * Willingness to continue using the product
  * Overall satisfaction
  Each item is scored from 0 (not satisfied at all) to 10 (completely satisfied). The total score ranges from 0 to 60. Higher scores indicate better satisfaction.
  Minimum Value: 0 Maximum Value: 60 Units of Measure: Points Meaning of Higher Scores: Better outcome (higher satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Pirawish Limlawan, D.D.S., Ph.D., Principal Investigator — Faculty of Dentistry, Chulalongkorn University

IPD SHARING:
Plan to Share IPD: No